CLINICAL TRIAL: NCT06736951
Title: Modifying the Inpatient Environment to Reduce the Incidence and Burden of Delirium Among Hospitalized Older Adults (≥70 Years).
Brief Title: Modifying the Inpatient Environment to Reduce Delirium in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Farhaan S. Vahidy (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Farhaan S. Vahidy, Adjunct Professor of Neurosurgery, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRO00037893
Record Dates: First submitted 2024-09-01; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Delirium; Sleep Hygiene
MeSH Terms: conditions — Delirium; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: This is a step-wedge cluster randomized controlled trials in which hospital units will cross over from control to intervention phase in a randomly assigned sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMSH (Multi-Modal Sleep Hygiene) Bundle (Experimental): We will implement an MMSH bundle, enhancing a previously reported sleep focused intervention, in order to increase quality/quantity of sleep during Z-time (i.e., 10pm to 5am) in our intervention units, subsequently mitigating the burden of delirium in hospitalized older adults. Our proposed intervention domains perfectly align with the expressed patient suggestions to improve patient experience. Sleep disruption issues were raised at similar rates across the age span suggesting our MMSH will positively impact patients of all ages, including those with lower risk of delirium. The intervention components are outlined below and a comparison to the current standard of care and the components that are relevant to the fidelity aspects of the study are highlighted in the table. The main focus of the sleep interventions will focus on Noise, Light, Staff-Patient Interactions, Daytime Activity and Medications.
  Interventions: Other: MMSH (Multi-Modal Sleep Hygiene) Bundle
- Standard of Care (No Intervention): This study arm reflects patients receiving standard of care treatment without any modification of in-hospital sleep environment

INTERVENTIONS:
Other: MMSH (Multi-Modal Sleep Hygiene) Bundle — Focus on Noise Reduce Noise Perception, Reduce Hallway Noise, Reduce Noise in Rooms Focus on Light Reduce Lights at Night, Increase Light in Day, Reduce Light Perception Focus on Staff-Patient Interactions Delirium Screening, Avoid Care Procedures at Night, Z-time Plan & Prep Focus on Daytime Activity Increased Mobility, Increase Patient Engagement Focus on Medications Pain Management, Medication Monitoring, Continue pharmacy protocols, Timing of Medications/Monitoring Labs
  Arms: MMSH (Multi-Modal Sleep Hygiene) Bundle

SUMMARY:
The overall goal is to reduce the incidence and burden of delirium, as measured by the delirium burden index (DBI) among hospitalized older adults (≥70 years), by modifying the inpatient environment to decrease its sleep antagonism. The investigators propose to implement a multi-modal sleep hygiene (MMSH) bundle, an enhancement of a previously reported sleep-focused intervention which had 88 - 100% compliance for intervention components, and reduced ICU delirium by 50%.

DETAILED DESCRIPTION:
The Investigators will implement the MMSH in a randomized step-wedge cluster design across 11 independent nursing units of 4 Methodist hospitals. While primarily focusing on the MMSH effectiveness, the investigators will conduct process evaluation to identify barriers and facilitators for MMSH implementation.

Specific Aim 1: Establish the comparative effectiveness of an in-hospital, MMSH towards reducing the rate of incident (hospital acquired) delirium (HAD) among older adults (age ≥ 70). The investigators will compare the rate of incident delirium between patients receiving the MMSH bundle in addition to the Standard of Care delirium screening and prevention protocol (SOC-DSPP), and those who are managed only under the SOC-DSPP. The SOC-DSPP through out all HM units includes twice daily deliruim screening with the 4AI. Outcome: The primary outcome is incident delirium (or HAD), determined by a positive 4AT, among patients who did not have delirium present on admission. The investigators hypothesize a 33% reduction in incident delirium among patients receiving the MMSH bundle.

Specific Aim 2: Establish the comparative effectiveness of an in-hospital, MMSH towards reducing delirium burden, as measured by DBI, among older adults (age ≥ 70), either with HAD or with D-POA. The investigators will compare the DBI between patients receiving the MMSH bundle in addition to the SOC-DSPP with that of those who were managed only under the SOC-DSPP. Outcome: The primary outcome is patient-level DBI [(number of positive 4AT screens)2/total number of 4AT screens)]. The DBI will be a non-zero positive fraction which is scale free because it accounts for the duration of observation by taking into consideration the total number of delirium assessments. Investigators hypothesize a 25% reduction in DBI among patients receiving the MMSH bundle.

Specific Aim 3: Evaluate the barriers and facilitators of implementing a MMSH bundle across community and academic hospitals and assess compliance with various MMSH bundle components. Outcomes: The outcomes are the reasons and factors that either promote or hinder implementation of the MMSH bundle. The investigators will also measure proportional compliance with each MMSH bundle component across the entire period implementation for all clusters (units).

Exploratory Aim: Compare sleep quality, as monitored by actigraphy, between patients receiving the MMSH bundle in addition to the SOC-DSPP with that of those who were managed under the SOC-DSPP only. Outcome: The outcomes are sleep duration, and frequency of awakenings during the hours of 10:00 pm and 5:00 am (i.e., Z-time) ,day to day variability and circadian rest-activity rhythm.

ELIGIBILITY:
Inclusion criteria:

* Non-critically ill patients (≥70 years)
* All sexes
* All races and ethnicities
* Admitted to the pre-specified clinical units which are part of the study

Exclusion criteria (applied during analysis):

* Patients with active alcohol or substance withdrawal.
* Patients with acute psychiatric illness
* Patients with initial admission to intensive care unit including requirement for mechanical ventilation.
* Patients present on a unit at the time of unit randomization

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10890 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence (cumulative or proportion) of hospital acquired delirium (HAD) among patients who did not have delirium present on admission (D-POA) | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Proportion of patients who develop HAD among those who did not have D-POA. D-POA is defined as 4AT positivity (at least one) during the first 48 hours of hospital admission. HAD is defined as 4AT positivity (at least one) after 48 hours of 4AT negatives.
Delirium Burden Index (DBI) among patients with either delirium present on admission or those who develop HAD | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Proportion of positive 4AT assessments (squared) among all 4AT assessments. Patient level metric of delirium burden. Scale free, non-zero number. [(#4AT+)2 / #Total 4AT]
Adherence to MMSH bundle components: Nighttime and Daytime | Starting from the date of randomization till the date of termination of the study assessments will be made twice weekly for each unit, up to 5 years
  Reported as frequency and proportion of patients among whom full implementation was possible. Frequency and proportion of adherence with individual bundle components.
Factors facilitating or impeding implementation of MMSH bundle | From the date of randomization assessments made up to 5 years
  Qualitative / thematic analysis of semi-structured focus groups with unit staff and PFAC stakeholders

SECONDARY OUTCOMES:
Resolution of delirium present on admission (D-POA) | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Proportion of D-POA patients who resolve delirium. Defined as no positive 4AT screens following 48-hours of hospitalization among those who were positive during first 48 hours
Delirium Assessment Positivity Rate | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Patient level indicator for the proportion of positive 4AT screen to the total number of 4AT screens for both D-POA and HAD patients
Length of Hospital Stay (days) | From the date of admission to the date of discharge or death, whichever comes first, up to 5 years
  Median (interquartile range) for number of days of hospitalization, compared between intervention and SOC patients
Delirium free days | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Among patients with either incident delirium or delirium present on admission, the number of days (24 hours periods) which were free of delirium (all negative 4AT screens).
In hospital mortality | Date of admission to the date of discharge or the date of death, which ever comes first, up to 5 years
  Proportion of patients experiencing in hospital mortality for intervention vs the SOC groups
Hospital discharge disposition | Date of admission to the date of discharge (for patients discharged alive), up to 5 years
  Favorable discharge disposition (home or rehab) vs. unfavorable disposition (SNF, LTAC, Nursing Home)
In Hospital complications | Date of admission to the date of discharge or death, whichever comes first, up to 5 years
  Pre-defined set of in-hospital complications (pneumonia, sepsis, UTI, DVT) will be tracked.
Need for higher level of care | Date of admission to the date of discharge or death, which ever comes first, up to 5 years
  Need for higher acuity care
Duration of daytime sleeping via actigraphy (non Z-time sleeping) | Baseline to Year 5
  Analysis of actigraphy data. Non - Z time sleep duration
Patient Experience | Baseline to Year 5
  HCAHPS scores in patients aged 65 and older by unit preintervention versus post intervention. The question used will be: "During this hospital stay, how often was the area around your room quiet at night?"
Mobilization/Daytime Activity | Date of admission to the date of discharge or death (which ever comes first), up to 5 years
  Mobility Dashboard data of Percentage of Patient Days per unit with Any Activity Documented in patients aged 70 or greater on the intervention unit
Sleep Quality for Actigraphy Patients | From the date of enrollment to the date of discharge or death, which ever comes first, assessed daily (for the daily survey), and assessed once post-discharge (for the post-discharge survey), up to 5 years
  Daily sleep quality survey and post-discharge sleep quality survey
Sleep quality for all enrolled patients | Date of admission to the date of discharge, or death, whichever comes first, assessed every other day, up to 5 years.
  Alternate day sleep quality survey for all enrolled patients (excluding actigraphy patients)
Incidence rate of hospital acquired delirium (HAD) among patients who did not have delirium present on admission (DPOA) | From the date of admission to the date of discharge or death, whichever comes first, outcome will be assessed at every 12 hours (twice in a 24 hour time period), up to 5 years
  Number of new cases of delirium (among those who were non-D-POA) per person-time.

OTHER OUTCOMES:
Duration of nighttime (10:00 pm to 5:00 am - 'Z-time') sleep time | Baseline to Year 5
  Analysis of actigraphy data.
Frequency of nocturnal (10:00 pm to 5:00 am - 'Z-time') awakenings | Baseline to Year 5
  Analysis of actigraphy data.

CONTACTS AND LOCATIONS:
Overall Officials: Farhaan Vahidy, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (5):
- United States (5):
  - Houston Methodist Baytown Hospital, Baytown, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Sugarland Hospital, Sugarland, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD is undecided.

REFERENCES:
- [Background] Patel J, Baldwin J, Bunting P, Laha S. The effect of a multicomponent multidisciplinary bundle of interventions on sleep and delirium in medical and surgical intensive care patients. Anaesthesia. 2014 Jun;69(6):540-9. doi: 10.1111/anae.12638. PMID 24813132
- See also: PCORI Webpage for Study — https://www.pcori.org/research-results/2023/improving-hospital-sleep-hygiene-prevent-and-curtail-delirium-among-older-adults